## **Informed Consent Form**



DocumentDate:30.08.2024

We invite you to participate in the project titled "The Effects of Different Dual Task Exercises on Motor and Cognitive Functions in Children with Mild Mental Retardation", conducted under the supervision of Associate Professor Dr. Yıldız ANALAY AKABABA at Istanbul University-Cerrahpaşa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. As a parent, if you agree to your child's participation in this study, you will be included in the voluntary group of the research. Information and data obtained from you and other participants will be used to reach a scientific conclusion. Before deciding whether to participate, it is important for you to understand why, how, and by what methods the study will be conducted, what is expected from you, and the benefits, risks, and discomforts that participation might bring.

Therefore, reading and understanding this form is important. If there is anything you do not understand or is unclear, please ask for clarification. Participation in the research is entirely voluntary. Only children whose parents voluntarily agree to participate will be included. You have the right not to participate or to withdraw at any time after enrolling. Please especially obtain information about the following topics related to the project:

- Nature of the project
- Purpose
- Contributions to science
- Procedures to be performed (e.g., blood draw, questionnaires)
- How it will be applied
- Which methods will be used (e.g., intravenous, interviews)
- Duration
- Approximate number of participants (if multi-center, total number of institutions and participants)
- Risks, possible adverse effects, and treatability

No fees will be charged to you or your child for any procedures within this project. This study will not affect your or your child's social security or other health insurance payments. Your and your child's identities will be kept confidential. However, if you wish, you will receive a report of the results obtained.

- ➤ This study is a master's thesis project.
- ➤ The title of the research is "The Effects of Different Dual Task Exercises on Motor and Cognitive Functions in Children with Mild Mental Retardation."
- ➤ The study will be conducted with children aged 8-12 diagnosed with mild mental retardation.
- The aim of this study is to investigate the effects of different dual task exercises on motor

and cognitive functions in children with mild mental retardation. The effects of exercises on cognitive function, walking, balance, and quality of life will be examined.

- ➤ After collecting demographic information, motor and cognitive functions will be assessed using questionnaires and scales at the beginning and after the 6-week exercise program, face-to-face.
- ➤ After all assessments, participants will be divided into three groups. Approximately 33 children aged 8-12 are planned to be included in the study.
- Two groups will perform dual task exercises; the first group will do motor-motor dual task exercises, the second group motor-cognitive dual task exercises. The third group will be given a home exercise program. Exercises will be applied twice a week for 6 weeks, each session lasting approximately 40 minutes.
- The assessments and exercises in the study are selected from scientific studies, will not cause discomfort, and do not involve expected risks.
- ➤ Throughout your participation, you are expected to attend all initial and final assessments and exercise sessions regularly.
- ➤ No fees will be charged, nor will you or your child be paid, for the assessments and exercise follow-up in this study.
- ➤ Participation is entirely voluntary. You can withdraw at any time without penalty or loss of benefits. Your and your child's identities will remain confidential, even if research results are published. Scientific results will be shared with you after the study. The data collector will be your contact person.
- The researcher may remove your child from the study if they do not attend exercise sessions, assessments, or if any health problems arise that affect treatment outcomes.
- ➤ If you encounter any problems during the research, you can contact Fzt. Melike Nur AKGÖĞ at (0)535 548 69 73.

"I have read all explanations in the informed consent form. I have been informed in writing and verbally by the data collector about the above-mentioned research topic and purpose. I voluntarily agree to participate in the study and understand that I can withdraw at any time, with or without reason."

Parent/Guardian Name and Surname:
Parent/Guardian Signature:
Parent/Guardian Contact Information:

Volunteer Name and Surname:

□ I agree to participate in the study

□ I do not agree to participate in the study

Researcher Name and Surname: Melike Nur AKGÖĞ

Researcher Signature:

Researcher Contact Information: (0)535 548 69 73